CLINICAL TRIAL: NCT02875639
Title: A Clinical Research of Qi Deficiency and Blood Stasis Syndrome (Different Disease With Syndrome)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhu Mingjun (Other)
Responsible Party: Sponsor-Investigator, Zhu Mingjun, Professor,chief physicians,the director of Henan University of Traditional Chinese Medicine, The First Affiliated Hospital of Henan University of Traditional Chinese Medicine
Organization: The First Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015CB554401
Record Dates: First submitted 2016-08-02; First posted 2016-08-23 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Ischemic Heart Failure
Keywords: Ischemic Heart Failure; coronary artery disease; qi deficiency and blood stasis
MeSH Terms: conditions — Coronary Artery Disease | interventions — buyang huanwu

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- tonifying qi group (Experimental): tonifying qi group:which treated by a kind of Chinese patent medicine (major components: Huangqi,Dangsheng,and so on)
  Interventions: Drug: Yiqi prescription; Drug: Placebo 1
- activating blood group (Experimental): which treated by a kind of Chinese patent medicine (major components: Honghua,Taoren,Danggui，and so on)
  Interventions: Drug: Huoxue prescription; Drug: Placebo 1
- qi and blood group (Experimental): which treated by a kind of Chinese patent medicine (major components: Huangqi,Dangsheng，Honghua,Taoren,Danggui，and so on)
  Interventions: Drug: Buyang huanwu decoction; Drug: Placebo 1
- QISHEN YIQI DRIPPING PILLS group (Active Comparator): which treated by a kind of Chinese patent medicine (major components: Huangqi,Dangsheng，and so on)
  Interventions: Drug: QISHEN YIQI DRIPPING PILLS; Drug: Placebo 2
- placebo group (Sham Comparator): which treated by the simulation of Chinese patent medicine (major components:excipient)
  Interventions: Drug: Placebo 1; Drug: Placebo 2

INTERVENTIONS:
Drug: Yiqi prescription
  Arms: tonifying qi group
Drug: Huoxue prescription
  Arms: activating blood group
Drug: Buyang huanwu decoction
  Arms: qi and blood group
Drug: QISHEN YIQI DRIPPING PILLS
  Arms: QISHEN YIQI DRIPPING PILLS group
Drug: Placebo 1 — Placebo 1：a drug which imitated QISHEN YIQI DRIPPING PILLS,but do not have active ingredient,just have the excipient.
  Arms: activating blood group; placebo group; qi and blood group; tonifying qi group
Drug: Placebo 2 — Placebo 2：a drug which imitated Buyang huanwu decoction,but do not have active ingredient,just have the excipient.
  Arms: QISHEN YIQI DRIPPING PILLS group; placebo group

SUMMARY:
The main purpose of this research is to reveal the curative effect mechanism of Yiqihuoxue prescription which treat the disease of qi deficiency and blood stasis. And at the same time this study also try to confirm yiqi huoxue fang qi deficiency blood stasis treatment of coronary heart disease (CHD) heart failure the curative effect and security.

DETAILED DESCRIPTION:
Modern research has shown that the main mechanism of the qi deficiency and blood stasis of coronary disease combined with cardiac failure is the disorder Nerve-endocrine-immune network mechanism, disorder of energy metabolism, blood coagulation/anticoagulation imbalances, vascular endothelial injury and the expression of inflammatory factors and cytokines disorder, etc. Some studies have identified that the Chinese traditional medicine of supplementing qi and activating blood circulation drugs could adjust the nerve - endocrine - immune network, improve endothelial function, improve ventricular remodeling, ameliorate heart function, alleviate the clinical symptoms, enhance the quality of life, and so on. This study by comparing the curative effect of Yi-Qi Formula, Huoxue prescription and two prescription of yiqi huoxue (buyang huanwu decoction and Qishen Yiqi Drop Pill) on improving energy metabolism, ameliorating heart function, adjusting the blood coagulation and the expression of cell adhesion factor, improving endothelial function, to reveal the curative effect mechanism of Yiqihuoxue prescription which treat the disease of qi deficiency and blood stasis, and confirm the TCM theory that "Qi and blood are correlated.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40 to 75;
2. Patients with ischemic heart failure： LVEF less than or equal to 45% measured by echocardiography in modified Simpson method
3. Qi deficiency and blood stasis syndrome;
4. New York Heart Association (NYHA) Class II to Ⅲ ;
5. Submitted informed consent

Exclusion Criteria:

1. Combin the pulmonary embolism, or acute coronary syndrome (acs) ,or acute cerebrovascular disease;
2. Combin other heart diseases: valvular heart disease, dilated cardiomyopathy, hypertension heart disease, pulmonary heart disease,congenital heart disease;
3. Hypertension and diabetes patients treated with drugs but not controlled within standard limit;
4. Severe hepatic and renal dysfunction, malnutrition, malignant tumour;
5. Active tuberculosis or rheumatoid diseases;
6. Nosohemia, organ transplantation,uremia;
7. Psychosis and drug abuse;
8. Allergic to the drugs or one component medicine of the drugs of this study ;
9. Participated in other trials within 1 month ;
10. Being pregnant, planning for pregnancy or breastfeeding;

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
N-terminal pronatriuretic peptide（NT-proBNP） | 0 month
N-terminal pronatriuretic peptide（NT-proBNP） | 3rd month
N-terminal pronatriuretic peptide（NT-proBNP） | 9th month

SECONDARY OUTCOMES:
Minnesota heart failure quality of life scale | 0,3rd,9th month
  baseline, 3 months after treatment and follow-up 6 months
sST2，Galectin3,PT,APTT,FBg,TT,TnT,CK,GLUT-1.GLUT-4,H-FABP | 0，3rd month
  the expression of these may be related to "Qi"
TXA2,PGI2,CD31,CD18,CD11b,R,K,MA | 0，3rd month
  the expression of these may be related to "Xue"
hs-CRP,IL-1β,IL-6,TNF-α,ICAM-1,VCAM-1,MCP-1,NO,ET-1 | 0，3rd month
  the expression of these may be related to "Mai"
Echocardiography | 0,3rd,9th month
  baseline, 3 months after treatment and follow-up 6 months
Cardiac magnetic resonance | 0，3rd month
  baseline, 3 months after treatment
Vascular ultrasound | 0，3rd month
  baseline, and after 3 months treatment
Endothelial function | 0，3rd month
  baseline, and after 3 months treatment
Cardiac function classification, NYHA | 0,1st,Sec,3rd,6th,9th,month
  baseline, 3 months after treatment and follow-up 6 months
ultrasonic cardiogram | 0,3rd,9th month
  baseline, 3 months after treatment and follow-up 6 months
6MWT distance | 0,3rd,9th month
  baseline, 3 months after treatment and follow-up 6 months
Traditional Chinese Medicine Syndrome Score Scale (TCMSSS) | 0,3rd,9th month
  baseline, 3 months after treatment and follow-up 6 months
blood and urine routine tests,liver and renal function tests,serum | 0,3rd,month
  safety evaluation
electrolytes,electrocardiogram (ECG) | 0,3rd,month
  safety evaluation
Composite endpoint | 1st,3rd,6th,9th, month
  all-cause death, frequency of emergency/re-admission to hospital due to HF, frequency of re-admission due to cardiovascular disease, acute coronary syndrome, severe arrhythmia, cardiac shock, revascularization, stroke, pulmonary embolism and peripheral vascular incidences, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Zhu M jun, Study Director — First affiliated hospital, Henan University of Traditional Chinese medicine; Wang Y xia, Principal Investigator — First affiliated hospital, Henan University of Traditional Chinese medicine; Li Bin, Principal Investigator — First affiliated hospital, Henan University of Traditional Chinese medicine
Locations (1):
- First affiliated hospital, Henan University of Traditional Chinese medicine, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] WRITING COMMITTEE MEMBERS; Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Drazner MH, Fonarow GC, Geraci SA, Horwich T, Januzzi JL, Johnson MR, Kasper EK, Levy WC, Masoudi FA, McBride PE, McMurray JJ, Mitchell JE, Peterson PN, Riegel B, Sam F, Stevenson LW, Tang WH, Tsai EJ, Wilkoff BL; American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. 2013 ACCF/AHA guideline for the management of heart failure: a report of the American College of Cardiology Foundation/American Heart Association Task Force on practice guidelines. Circulation. 2013 Oct 15;128(16):e240-327. doi: 10.1161/CIR.0b013e31829e8776. Epub 2013 Jun 5. No abstract available. PMID 23741058
- [Derived] Zhao Z, Jin X, Li Y, Wang X, Cui Y, Zhang B, Kang Y, Zhang G, Chu Q, Zhang J. Efficacy and safety of fospropofol disodium sedation for same-day bidirectional endoscopy in elderly patients: protocol for a prospective, single-center, randomized, double-blind, non-inferiority trial. Front Pharmacol. 2024 Aug 8;15:1378081. doi: 10.3389/fphar.2024.1378081. eCollection 2024. PMID 39175547